CLINICAL TRIAL: NCT00775515
Title: Laparoscopic Prostatectomy for Chronic Prostatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Krongrad Institute (Other)
Responsible Party: ARNON KRONGRAD,M.D., THE KRONGRAD INSTITUTE
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20081635
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Prostatitis; Chronic Prostatitis With Chronic Pelvic Pain Syndrome
Keywords: chronic; prostatitis; prostate; pain; pelvic; pelvis; inflamation
MeSH Terms: conditions — Prostatitis; Bronchiolitis Obliterans Syndrome; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one (Experimental): laparoscopic prostatectomy
  Interventions: Procedure: laparoscopic prostatectomy

INTERVENTIONS:
Procedure: laparoscopic prostatectomy — laparoscopic prostatectomy
  Other Names: laparoscopic radical prostatectomy; minimally invasive prostate surgery

SUMMARY:
Prostatitis is an inflammation of the prostate, an pelvic organ of men. Prostatitis can cause great discomfort which varies but can include pelvic pain, pelvic pressure, a vague sense of discomfort, a feeling of malaise and fatigue, fever, burning on urination, pain on reaching orgasm, and bleeding.

In many men the symptoms of prostatitis can be chronic. It is estimated that in the United States chronic prostatitis is responsible for as many as two million doctor visits a year. The disease can be ruinous, interfering with work, intimacy, and other things.

The causes of chronic prostatitis are not understood. The treatments commonly used, including antibiotics and prostate massage, work poorly. We now have evidence that laparoscopic prostatectomy can eliminate the misery of chronic prostatitis. This trial aims to quantify and better characterize the effect of laparoscopic prostatectomy on the symptoms of chronic prostatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 and greater
* NIH-CPSI score of 25 and higher
* Symptom duration of at least one year
* Failed treatment with antibiotics and/or other medications

Exclusion Criteria:

* Inability to tolerate Anesthesia
* Inability to speak any English

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
NHI CPSI (chronic prostatitis symptom index) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Krongrad, MD, Principal Investigator — The Krongrad Institute
Locations (1):
- The Krongrad Institute, Aventura, Florida, United States

REFERENCES:
- [Result] Krongrad A, Lai S: Laparoscopic Prostatectomy for Severely Symptomatic, Treatment-Refractory Chronic Prostatitis: Preliminary Observations from an Ongoing Phase II Clinical Trial. UroToday Int J. 2011 Apr;4(2) http://bit.ly/iLkwht
- See also: Get More Information and Download Informed Consent — http://ProstatitisSurgery.com